CLINICAL TRIAL: NCT00906997
Title: Colorectal Cancer Screening in Average-risk Population: a Multicenter, Randomized Control Trial Comparing Immunochemical Fecal Occult Blood Testing Versus Colonoscopy.
Brief Title: Colorectal Cancer Screening in Average-risk Population: Immunochemical Fecal Occult Blood Testing Versus Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundacion Cientifica de la Asociacion Española contra el Cancer (Unknown); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Antoni Castells, Co-principal investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: COLONPREV
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Colorectal Neoplasm
Keywords: Colorectal cancer; Screening; Prevention; Fecal occult blood test; Colonoscopy; Colorectal neoplasm; Randomized clinical trial
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fecal occult blood testing (Active Comparator): Fecal immunochemical testing biennially
  Interventions: Procedure: Immunochemical fecal occult blood test
- Colonoscopy (Active Comparator): Colonoscopy one time
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Immunochemical fecal occult blood test — Biennial, without diet restriction, 1 stool sample. Positive cut-off level: 75 ng/ml.
  Arms: Fecal occult blood testing
Procedure: Colonoscopy — Every 10 years, with sedation.
  Arms: Colonoscopy

SUMMARY:
Aims:

1. To compare the efficacy of biennial immunochemical fecal occult blood test (iFOBT) versus colonoscopy every 10 years for the reduction of colorectal cancer-related mortality at 10 years in average-risk population.
2. To determine the compliance and complications associated with both strategies.

Methods: Multicenter, randomized, controlled study in 8 Spanish regions (Aragón, Canarias, Catalunya, Euskadi, Galicia, Madrid, Murcia and Valencia).

Study groups:

* Group I: iFOBT (OC Sensor®) in one stool sample, followed by colonoscopy when a positive result.
* Group II: colonoscopy.

Sample-size calculation: 27,749 subjects in each study group (total: 55,498).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 50-69 years

Exclusion Criteria:

* Personal history of colorectal cancer, colorectal adenoma, colorectal polyposis, or inflammatory bowel disease
* Family history of colorectal polyposis, Lynch syndrome or familial colorectal cancer (2 or more first-degree relatives diagnosed with colorectal cancer or one first-degree relative diagnosed with colorectal cancer before the age of 60)
* Severe comorbidity
* Previous total colectomy
* Not signed informed consent to participate

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55498 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer-related mortality | 10 years

SECONDARY OUTCOMES:
Compliance rate | 2 years
Complication rate | 10 years
Colorectal cancer incidence | 15 years
Adherence rate | 10 years
Advanced colorectal neoplasm detection rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Castells, MD, Principal Investigator — Hospital Clínic, Barcelona, Spain; Enrique Quintero, MD, Principal Investigator — Hospital Universitario de Canarias, Tenerife, Spain
Locations (8):
- Spain (8):
  - Hospital del Mar, Barcelona
  - Hospital Clínico, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Meixoeiro, Ourense
  - Hospital de Donosti, San Sebastián
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Comunidad Valencia, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Castells A, Quintero E, Bujanda L, Castan-Cameo S, Cubiella J, Diaz-Tasende J, Lanas A, Ono A, Serra-Burriel M, Frias-Arrocha E, Hernandez C, Jover R, Andreu M, Carballo F, Morillas JD, Salas D, Almazan R, Alonso-Abreu I, Banales JM, Hernandez V, Portillo I, Vanaclocha-Espi M, de la Vega M; COLONPREV study investigators. Effect of invitation to colonoscopy versus faecal immunochemical test screening on colorectal cancer mortality (COLONPREV): a pragmatic, randomised, controlled, non-inferiority trial. Lancet. 2025 Apr 12;405(10486):1231-1239. doi: 10.1016/S0140-6736(25)00145-X. Epub 2025 Mar 27. PMID 40158525
- [Derived] Shaukat A, Kahi CJ, Burke CA, Rabeneck L, Sauer BG, Rex DK. ACG Clinical Guidelines: Colorectal Cancer Screening 2021. Am J Gastroenterol. 2021 Mar 1;116(3):458-479. doi: 10.14309/ajg.0000000000001122. PMID 33657038
- [Derived] Salas D, Vanaclocha M, Ibanez J, Molina-Barcelo A, Hernandez V, Cubiella J, Zubizarreta R, Andreu M, Hernandez C, Perez-Riquelme F, Cruzado J, Carballo F, Bujanda L, Sarasqueta C, Portillo I, de la Vega-Prieto M, Morillas JD, Valentin V, Lanas A, Quintero E, Castells A. Participation and detection rates by age and sex for colonoscopy versus fecal immunochemical testing in colorectal cancer screening. Cancer Causes Control. 2014 Aug;25(8):985-97. doi: 10.1007/s10552-014-0398-y. Epub 2014 May 24. PMID 24859111
- [Derived] Castells A, Quintero E, Alvarez C, Bujanda L, Cubiella J, Salas D, Lanas A, Carballo F, Morillas JD, Hernandez C, Jover R, Hijona E, Portillo I, Enriquez-Navascues JM, Hernandez V, Martinez-Turnes A, Menendez-Villalva C, Gonzalez-Mao C, Sala T, Ponce M, Andres M, Teruel G, Peris A, Sopena F, Gonzalez-Rubio F, Seoane-Urgorri A, Grau J, Serradesanferm A, Pozo A, Pellise M, Balaguer F, Ono A, Cruzado J, Perez-Riquelme F, Alonso-Abreu I, Carrillo-Palau M, de la Vega-Prieto M, Iglesias R, Amador J, Blanco JM, Sastre R, Ferrandiz J, Gonzalez-Hernandez MJ, Andreu M, Bessa X; COLONPREV Study Investigators. Rate of detection of advanced neoplasms in proximal colon by simulated sigmoidoscopy vs fecal immunochemical tests. Clin Gastroenterol Hepatol. 2014 Oct;12(10):1708-16.e4. doi: 10.1016/j.cgh.2014.03.022. Epub 2014 Mar 27. PMID 24681078
- [Derived] Hernandez V, Cubiella J, Gonzalez-Mao MC, Iglesias F, Rivera C, Iglesias MB, Cid L, Castro I, de Castro L, Vega P, Hermo JA, Macenlle R, Martinez-Turnes A, Martinez-Ares D, Estevez P, Cid E, Vidal MC, Lopez-Martinez A, Hijona E, Herreros-Villanueva M, Bujanda L, Rodriguez-Prada JI; COLONPREV Study Investigators. Fecal immunochemical test accuracy in average-risk colorectal cancer screening. World J Gastroenterol. 2014 Jan 28;20(4):1038-47. doi: 10.3748/wjg.v20.i4.1038. PMID 24574776
- [Derived] Bujanda L, Lanas A, Quintero E, Castells A, Sarasqueta C, Cubiella J, Hernandez V, Morillas JD, Perez-Fernandez T, Salas D, Andreu M, Carballo F, Bessa X, Cosme A, Jover R; COLONPREV Study Investigators. Effect of aspirin and antiplatelet drugs on the outcome of the fecal immunochemical test. Mayo Clin Proc. 2013 Jul;88(7):683-9. doi: 10.1016/j.mayocp.2013.04.016. Epub 2013 Jun 7. PMID 23751980
- [Derived] Quintero E, Castells A, Bujanda L, Cubiella J, Salas D, Lanas A, Andreu M, Carballo F, Morillas JD, Hernandez C, Jover R, Montalvo I, Arenas J, Laredo E, Hernandez V, Iglesias F, Cid E, Zubizarreta R, Sala T, Ponce M, Andres M, Teruel G, Peris A, Roncales MP, Polo-Tomas M, Bessa X, Ferrer-Armengou O, Grau J, Serradesanferm A, Ono A, Cruzado J, Perez-Riquelme F, Alonso-Abreu I, de la Vega-Prieto M, Reyes-Melian JM, Cacho G, Diaz-Tasende J, Herreros-de-Tejada A, Poves C, Santander C, Gonzalez-Navarro A; COLONPREV Study Investigators. Colonoscopy versus fecal immunochemical testing in colorectal-cancer screening. N Engl J Med. 2012 Feb 23;366(8):697-706. doi: 10.1056/NEJMoa1108895. PMID 22356323
- See also: Webpage of the Spanish Gastroenterological Association, which endorses COLONPREV trial — http://www.aegastro.es

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT00906997/Prot_SAP_000.pdf